CLINICAL TRIAL: NCT04162743
Title: The Effect of Trazodone on the Severity of Obstructive Sleep Apnea in Insomnic Stroke Patients With Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHEN,CHUNG YAO, doctor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMRPG2I0021
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Sleep Apnea Syndromes; Cerebral Infarction
MeSH Terms: conditions — Sleep Apnea Syndromes; Cerebral Infarction | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trazodone (Active Comparator): take trazodone 100mg hs
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): take placebo pill hs
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Trazodone — take trazodone 100mg before polysomnography
  Arms: Trazodone
Drug: Placebo oral tablet — take placebo oral tablet before polysomnography
  Arms: Placebo

SUMMARY:
The investigators hypothesize that trazodone does not worse nocturnal oxygen saturation in insomnic ischemic stroke patients with obstructive sleep apnea (OSA) and depression and has beneficial effect in selected stroke patients with low arousal threshold phenotype OSA.

ELIGIBILITY:
Inclusion Criteria:

* Insomnic ischemic stroke patients with OSA and depression.

Exclusion Criteria:

* unclear consciousness, unstable vital sign or neurologic sign, unstable medical conditions such as delirium, active infection, evidence of overt congestive cardiac failure, liver dysfunction with ascites, thyroid disease, end-stage-renal-disease receiving dialysis.
* overnight mean oxygen saturation (SaO2) nadir is ≤ 70% at baseline
* take monoamine oxidase inhibitors (MAOI), any medication that may affect breathing, sleep, or muscle activity
* any known allergy to trazodone
* sleep disorder other than OSA (e.g., periodic leg movement syndrome, restless legs syndrome, central sleep apnea/Cheyne-Stokes respiration).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
nocturnal oxygen saturation | the polysomnography study night before take drug
  mean and minimum oxyhemoglobin saturation (%) detected by pulse oximetry during polysomnography study
Sleep apnea severity index | the polysomnography study night before take drug
  apnea-hypopnea index, desaturation index according to The American Academy of Sleep Medicine (AASM) scoring manual version 2.0.3: Obstructive apnea: no airflow >= 10 s with respiratory effort (per hour of time); central apnea: no airflow without respiratory effort (per hour of time). Hypopnea: airflow decrease >30% lasting >= 10 s, followed by either oxygen desaturation > 3% or EEG arousal (per hour of time). The desaturation index: number of desaturations per hour of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen CY, Chen CL, Yu CC. Trazodone improves obstructive sleep apnea after ischemic stroke: a randomized, double-blind, placebo-controlled, crossover pilot study. J Neurol. 2021 Aug;268(8):2951-2960. doi: 10.1007/s00415-021-10480-2. Epub 2021 Feb 24. PMID 33625584